CLINICAL TRIAL: NCT00520598
Title: A Phase IIa Randomized, Double-Blind Controlled With Gardasil, Clinical Trial to Study theTolerability and Immunogenicity of V505 (a Multivalent Human Papilloma Virus [HPV] L1 Virus Like Particle [VLP] Vaccine) in Healthy 16 to 26 Year Old Women
Brief Title: Broad Spectrum HPV (Human Papillomavirus) Vaccine in 16 to 26 Year Old Women (V505-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V505-001; 2007_567
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Cervical Cancer; Vulvar Cancer; Vaginal Cancer; Genital Warts; Human Papillomavirus Infection
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata; Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Active Comparator): Arm 1: 0.5 ml injection of Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine as 3 dose regimen.
  Interventions: Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant
- 2 (Experimental): Arm 2: 0.5 ml injection of V505 formulation 1 as 3 dose regimen.
  Interventions: Biological: Comparator: V505 formulation 1
- 3 (Experimental): Arm 3: 0.5 ml injection of V505 formulation 2 as 3 dose regimen
  Interventions: Drug: Comparator: V505 formulation 2
- 4 (Experimental): Arm 4: 0.5 ml injection of V505 formulation 2 as 2 dose regimen and 1 Pbo injection
  Interventions: Drug: Comparator: V505 formulation 2; Biological: Comparator: Placebo (unspecified)
- 5 (Experimental): Arm 5: 0.5 ml injection of V505 formulation 3 as 2 dose regimen and 1 Pbo injection
  Interventions: Biological: Comparator: V505 formulation 3; Biological: Comparator: Placebo (unspecified)

INTERVENTIONS:
Biological: Comparator: V505 formulation 1 — 0.5 ml injection of V505 formulation 1 as 3 dose regimen at Day 1, Month 2 and Month 6.
  Arms: 2
Drug: Comparator: V505 formulation 2 — 0.5 ml injection of V505 formulation 2 as 3 dose regimen at Day 1, Month 2 and Month 6.
  Arms: 3
Drug: Comparator: V505 formulation 2 — 0.5 ml injection of V505 formulation 2 as 2 dose regimen at Day 1 and Month 6.
  Arms: 4
Biological: Comparator: V505 formulation 3 — 0.5 ml injection of V505 formulation 3 as 2 dose regimen at Day 1 and Month 6.
  Arms: 5
Biological: Comparator: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant — 0.5 ml injection of Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine as 3 dose regimen at Day 1, Month 2 and Month 6.
  Arms: 1
Biological: Comparator: Placebo (unspecified) — 0.5 ml injection of placebo to V505 as a 1 dose regimen at Month 2.
  Arms: 4; 5

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of V505 in comparison to GARDASIL (TM)

ELIGIBILITY:
Inclusion Criteria:

* Female between 16 to 26 years old
* Has never had Pap testing or have only had normal Pap test results
* Lifetime history of 0 to 4 sexual partners

Exclusion Criteria:

* History of an abnormal cervical biopsy result; History of a positive test for HPV; History of external genital/vaginal warts; Currently a user of any illegal drugs or an alcohol abuser
* History of severe allergic reaction that required medical attention
* Are pregnant
* Received a marketed HPV vaccine
* Currently enrolled in a clinical trial
* Currently has (or has a history of) certain medical conditions or is currently taking or has taken certain medications (details will be discussed at time of consent)

Ages: 16 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 511 (Actual)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) to HPV types contained in the vaccines administered in a 3-dose regimen | 4 weeks post dose 3

SECONDARY OUTCOMES:
Geometric mean titers (GMTs) to HPV types contained in the vaccines administered in a 2-dose regimen | 4 weeks post dose 2

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263